CLINICAL TRIAL: NCT03825419
Title: Muscle Assessment in Stroke Study (MASS): Detection of Muscle Loss in Acute Stroke Patients Who Need Enteral Nutrition
Brief Title: Detection of Muscle Loss in Acute Stroke Patients Who Need Enteral Nutrition (MASS)
Acronym: MASS
Status: Completed | Type: Observational
Sponsor: Turkish Stroke Research and Clinical Trials Network (Network)
Collaborators: Abbott Nutrition (Industry); Klinar CRO (Other); Turkish Neurological Society (Unknown)
Responsible Party: Principal Investigator, Ethem Murat Arsava, Prof.Dr., Turkish Stroke Research and Clinical Trials Network
Other Study IDs: MASS
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke, Acute, Neurocritical Care, Nutrition, Sarcopenia
MeSH Terms: conditions — Ischemic Stroke; Stroke; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The degree of muscle loss over the course of inpatient stay will be evaluated in patients with a diagnosis of acute ischemic stroke admitted to Neurocritical Care Units and necessitating enteral nutrition.

DETAILED DESCRIPTION:
This study is a multicenter, prospective observational study. The study period is 12 months. There are no investigational products to be followed or used in the study.

Demographic data, stroke subtype, lesion localization, anthropometric measures will be recorded. Muscle in three different anatomical sites will be measured by CT following admission in patients included in the study.

For anthropometric measurements, height, body weight, body mass index, waist circumference, triceps skin thickness and calf circumference values will be used.

The muscle mass will be measured from the paraspinal muscles at the L3 vertebra level and from the muscles around the humerus and femur on the non-paralytic side of the extremities by CT.

All patients will receive standard enteral nutritional support with a standardized calorie and protein-based protocol recommended by international guidelines. The choice of the commercial enteral product will be left to the investigator, without any encouragement or restriction for use of any commercial product.

The enteral nutrition protocol will be implemented as follows;

* Nasogastric or nasojejunal access
* Continuous infusion
* Targeted daily calories - 25-30 kcal / kg
* Targeted daily protein - 1.2-1.5 gr / kg
* 20 ml / h initial infusion rate
* Increase infusion rate by 10-20 ml / h in 8-12 hours
* Targeted calorie-protein requirement will be reached at the end of 72 hours.

Patients will continue their routine follow-up in the neurology intensive care unit / stroke unit / neurology department. Daily enteral nutrition dose, complications attributed to enteral nutrition and systemic comorbidities will be recorded. Anthropometric measurements and muscle mass measurements with CT at three different locations will be repeated at the end of the second week (14 days ± 3 days) .

The study will evaluate whether or not muscle mass develops 14 days after acute ischemic stroke. The end points of the study is deterioration of anthropometric measurements and loss of muscle mass demonstrated by CT at follow up. The differences between patients with and without muscle loss will be assessed from the the aspects of demographic characteristics, ischemic stroke subtype, comorbidities and the success attained in reaching enteral nutritional goals.

ELIGIBILITY:
Inclusion Criteria:

Patients to be included in this study are required to meet all of the following inclusion criteria:

* Acute ischemic stroke
* Admission within first 24 hours after symptom onset
* Admission NIHSS score > 8
* Being unable to walk
* Need for enteral tube feeding due to problems with consciousness or dysphagia

Exclusion Criteria:

Patients with any of the following exclusion criteria can not be included in the study:

* Retained ability for oral feeding
* Known muscle disease, neuropathy, neuromuscular junction disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of acute ischemic stroke admitted to Neurocritical Care Units for whom enteral nutrition is indicated
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass | 14 days
  Comparison of anthropometric measurements and CT based muscle mass measurements obtained at admission and at day 14 (± 3 days)

CONTACTS AND LOCATIONS:
Locations (10):
- Turkey (Türkiye) (10):
  - Ankara University Faculty of Medicine, Ankara
  - Gazi University Faculty Of Medicine, Ankara
  - Hacettepe University Faculty of Medicine, Ankara
  - Eskişehir Osmangazi Faculty of Medicine, Eskişehir
  - Gaziantep University Faculty of Medicine, Gaziantep
  - İstanbul Şişli Hamidiye Etfal Training and Research Hospital, Istanbul
  - Dokuz Eylül University Faculty of Medicine, Izmir
  - Ege University Faculty of Medicine, Izmir
  - İzmir Katip Çelebi University Atatürk Training and Research Hospital, Izmir
  - Ondokuz Mayıs University Faculty of Medicine, Samsun

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shiraishi A, Yoshimura Y, Wakabayashi H, Tsuji Y. Prevalence of stroke-related sarcopenia and its association with poor oral status in post-acute stroke patients: Implications for oral sarcopenia. Clin Nutr. 2018 Feb;37(1):204-207. doi: 10.1016/j.clnu.2016.12.002. Epub 2016 Dec 10. PMID 28017450
- [Background] Scherbakov N, Sandek A, Doehner W. Stroke-related sarcopenia: specific characteristics. J Am Med Dir Assoc. 2015 Apr;16(4):272-6. doi: 10.1016/j.jamda.2014.12.007. Epub 2015 Feb 10. PMID 25676847
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Coelen RJ, Wiggers JK, Nio CY, Besselink MG, Busch OR, Gouma DJ, van Gulik TM. Preoperative computed tomography assessment of skeletal muscle mass is valuable in predicting outcomes following hepatectomy for perihilar cholangiocarcinoma. HPB (Oxford). 2015 Jun;17(6):520-8. doi: 10.1111/hpb.12394. Epub 2015 Feb 28. PMID 25726722
- [Derived] Gungor L, Arsava EM, Guler A, Togay Isikay C, Aykac O, Batur Caglayan HZ, Kozak HH, Aydingoz U, Topcuoglu MA; MASS investigators. Determinants of in-hospital muscle loss in acute ischemic stroke - Results of the Muscle Assessment in Stroke Study (MASS). Clin Nutr. 2023 Mar;42(3):431-439. doi: 10.1016/j.clnu.2023.01.017. Epub 2023 Feb 3. PMID 36805095